CLINICAL TRIAL: NCT00433160
Title: Efficacy and Safety of LY333334 in Japanese Patients With Osteoporosis
Brief Title: Phase 3 Clinical Trial of Teriparatide in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10494; B3D-JE-GHDB (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Results first posted 2009-09-30 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Teriparatide (Experimental): 20 micrograms for 104 weeks
  Interventions: Drug: Teriparatide
- Placebo (Placebo Comparator): Placebo for 52 weeks. After 52 weeks, all patients on placebo can receive 20 micrograms teriparatide for 52 weeks
  Interventions: Drug: Teriparatide; Drug: Placebo

INTERVENTIONS:
Drug: Teriparatide — daily, subcutaneous
  Other Names: LY333334; Forteo; Forsteo
Drug: Placebo — daily, subcutaneous
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of teriparatide based on measurements of bone mineral density at lumbar spine

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients diagnosed with osteoporosis
* Aged 55 or older
* Patients who are at high risk for fracture

Exclusion Criteria:

* History of metabolic bone disorders other than primary osteoporosis
* History of malignant neoplasm in the 5 years, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitively treated.
* Severe or chronically disabling conditions other than osteoporosis

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- Japan (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Numakunai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shimane
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tottori

REFERENCES:
- [Result] Miyauchi A, Matsumoto T, Sugimoto T, Tsujimoto M, Warner MR, Nakamura T. Effects of teriparatide on bone mineral density and bone turnover markers in Japanese subjects with osteoporosis at high risk of fracture in a 24-month clinical study: 12-month, randomized, placebo-controlled, double-blind and 12-month open-label phases. Bone. 2010 Sep;47(3):493-502. doi: 10.1016/j.bone.2010.05.022. Epub 2010 May 24. PMID 20580870
- [Derived] Yamamoto T, Tsujimoto M, Sowa H. Safety of daily teriparatide treatment: a post hoc analysis of a Phase III study to investigate the possible association of teriparatide treatment with calcium homeostasis in patients with serum procollagen type I N-terminal propeptide elevation. Clin Interv Aging. 2015 Jul 6;10:1101-9. doi: 10.2147/CIA.S83549. eCollection 2015. PMID 26185429
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Results from 4 patients aren't included in baseline and outcomes: 3 (2 placebo and 1 teriparatide) didn't receive study drug; 1 (placebo) had a significant good clinical practice issue of receiving study drug assigned to another patient.
Period: 52-Week Double-Blind (DB) Period
Arm/Group | Teriparatide | Placebo
Started | 137 | 70
Received Treatment | 136 | 68
Completed | 120 | 60
Not Completed | 17 | 10
Not completed — Adverse Event | 6 | 2
Not completed — Death | 0 | 0
Not completed — Lost to Follow-up | 0 | 0
Not completed — Entry Criteria Exclusion | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Physician Decision | 4 | 2
Not completed — Sponsor Decision | 0 | 0
Not completed — Lack of Efficacy | 1 | 2
Period: 76 Weeks, 24-Week Open Label (OL) Period
Arm/Group | Teriparatide | Placebo
Started | 119 (One participant did not continue to first OL period due to adverse event after completing DB period.) | 59 (One participant did not continue to first OL period due to adverse event after completing DB period.)
Received Treatment | 119 | 59
Completed | 113 | 55
Not Completed | 6 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Lack of Efficacy | 0 | 1
Period: 104 Weeks, 28-Week OL Period
Arm/Group | Teriparatide | Placebo
Started | 102 (Eleven participants withdrew at end of first OL period and did not continue on to second OL period.) | 50 (Five participants withdrew at end of first OL period and did not continue on to second OL period.)
Received Treatment | 102 | 50
Completed | 92 | 47
Not Completed | 10 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Placebo | Total
Number analyzed (Participants) | 136 | 67 | 203
Age Continuous [Mean (Standard Deviation); unit: years] | 69.2 (6.3) | 70.4 (5.4) | 69.6 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 62 | 189
  Male | 9 | 5 | 14
Region of Enrollment [Number; unit: participants]
  Japan | 136 | 67 | 203
Alcohol Consumption [Number; unit: participants]
  No | 99 | 51 | 150
  Yes | 37 | 16 | 53
Number of Previous Vertebral Fractures [Number; unit: participants]
  0 Fractures | 82 | 38 | 120
  1 Fracture | 35 | 16 | 51
  2 Fractures | 10 | 8 | 18
  3 Fractures | 3 | 3 | 6
  4 Fractures | 4 | 1 | 5
  5 or More Fractures | 2 | 1 | 3
Previous Osteoporosis Drug Use [Number; unit: participants]
  No | 86 | 44 | 130
  Yes | 50 | 23 | 73
Smoking History [Number; unit: participants]
  Non-Smoker | 114 | 53 | 167
  Past Smoker | 6 | 9 | 15
  Current Smoker | 16 | 5 | 21
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared (kg/m^2).
  kilograms per square meter (kg/m^2) | 21.58 (3.03) | 22.24 (3.34) | 21.80 (3.15)
Bone Mineral Density (BMD) Total Spine [Mean (Standard Deviation); unit: grams per square centimeter (g/cm^2)] | 0.6153 (0.0701) | 0.6123 (0.0780) | 0.6143 (0.0726)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 150.40 (5.97) | 150.30 (5.74) | 150.36 (5.89)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 48.74 (6.83) | 50.25 (8.10) | 49.24 (7.29)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Bone Mineral Density at Lumbar Spine (L2-L4)
Description: Percent change in bone mineral density (BMD) at lumbar spine (L2-L4) from baseline to the last measurement point.
Time Frame: Baseline to 52 weeks
Population: Number of randomized participants with at least one dose of study drug and at least one post-treatment measurement.
Measure: Mean (Standard Deviation); unit: percent change in BMD
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 131 | 63
percent change in BMD
  Percent Change to Last Measurement Point | 9.82 (5.36) | 0.04 (4.34)
Statistical Analysis 1: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in bone mineral density at lumbar spine (L2-L4) after 52-week treatment between the two treatment groups; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Percent Change to Last Measurement Point. No adjustments for multiplicity was performed

2. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) at Lumbar Spine (L1-L4)
Description: Percent change in bone mineral density at lumbar spine (L1-L4) from baseline to the last measurement point.
Time Frame: Baseline to 52 Weeks
Population: Number of randomized participants who received at least one dose of study drug and with at least one post-treatment measurement.
Measure: Mean (Standard Deviation); unit: percent change in BMD
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 131 | 63
percent change in BMD
  Percent Change to Last Measurement Point | 10.23 (5.74) | 0.11 (4.42)

3. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) at Total Hip
Description: Percent change in bone mineral density (BMD) at total hip from baseline to the last measurement point.
Time Frame: Baseline to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in BMD
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 130 | 62
percent change in BMD
  Percent Change to Last Measurement Point | 2.66 (4.22) | -0.22 (3.38)

4. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) at Femoral Neck
Description: Percent change in bone mineral density at femoral neck from baseline to the last measurement point.
Time Frame: Baseline to 52 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in BMD
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 130 | 62
percent change in BMD
  Percent Change to Last Measurement Point | 2.24 (6.01) | 0.46 (3.89)

5. Secondary Outcome: Percent Change in Biochemical Markers of Bone Metabolism - Serum Procollagen I N-terminal Propeptide (PINP)
Description: Percent change in serum procollagen I N-terminal propeptide (PINP) from baseline to the individual visits and last measurement point.
Time Frame: Baseline to Weeks 4, 12, 24, and 52
Population: Number of randomized participants with at least one dose of study drug and with at least one post-treatment measurement.
Measure: Mean (Standard Deviation); unit: percent change in PINP
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 136 | 67
percent change in PINP
  Percent Change to Week 4 (n=136, n=66) | 90.67 (49.85) | -9.58 (14.39)
  Percent Change to Week 12 (n=131, n=64) | 89.58 (66.58) | -16.89 (17.35)
  Percent Change to Week 24 (n=127, n=61) | 114.12 (112.04) | -19.10 (29.17)
  Percent Change to Week 52 (n=121, n=60) | 116.11 (139.72) | -14.18 (29.02)
  Percent Change to Last Measurement (n=136,n=66) | 111.74 (134.38) | -13.82 (28.42)
Statistical Analysis 1: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in PINP after 4-week treatment between the two treatment groups; Test type: Superiority or Other; p < 0.001, Wilcoxon's Rank Sum Test — P-value for Percent Change to Week 4. No adjustment for multiplicity was performed
Statistical Analysis 2: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in PINP after 12-week treatment between the two treatment groups; Test type: Superiority or Other; p < 0.001, Wilcoxon's Rank Sum Test — P-value for Percent Change to Week 12. No adjustment for multiplicity was performed
Statistical Analysis 3: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in PINP after 24-week treatment between the two treatment groups; Test type: Superiority or Other; p < 0.001, Wilcoxon's Rank Sum Test — P-value for Percent Change to Week 24. No adjustment for multiplicity was performed
Statistical Analysis 4: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in PINP after 52-week treatment between the two treatment groups; Test type: Superiority or Other; p < 0.001, Wilcoxon's Rank Sum Test — P-value for Percent Change to Week 52. No adjustment for multiplicity was performed
Statistical Analysis 5: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in PINP from baseline to the last measurement point between the two treatment groups; Test type: Superiority or Other; p < 0.001, Wilcoxon's Rank Sum Test — P-value for Percent Change to Last Measurement. No adjustment for multiplicity was performed

6. Secondary Outcome: Percent Change in Biochemical Markers of Bone Metabolism - Serum Bone-specific Alkaline Phosphatase (BAP)
Description: Percent change in serum bone-specific alkaline phosphatase (BAP) from baseline to the individual visits and last measurement point.
Time Frame: Baseline to Weeks 4, 12, 24, 52
Population: Number of randomized participants with at least one dose of study drug and with at least one post-treatment measurement.
Measure: Mean (Standard Deviation); unit: percent change in BAP
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 136 | 67
percent change in BAP
  Percent Change to Week 4 (n=135, n=66) | 3.74 (37.86) | -9.63 (33.62)
  Percent Change to Week 12 (n=131, n=62) | 3.23 (49.05) | -16.97 (40.54)
  Percent Change to Week 24 (n=127, n=60) | -4.60 (43.44) | -28.46 (23.81)
  Percent Change to Week 52 (n=120, n=59) | -17.69 (58.12) | -32.24 (46.95)
  Percent Change to Last Measurement (n=136, n=66) | -17.32 (56.06) | -28.34 (46.96)
Statistical Analysis 1: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in BAP after 4-week treatment between the two treatment groups; Test type: Superiority or Other; p < 0.001, Wilcoxon's Rank Sum Test — P-value for Percent Change to Week 4. No adjustment for multiplicity was performed
Statistical Analysis 2: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in BAP after 12-week treatment between the two treatment groups; Test type: Superiority or Other; p < 0.001, Wilcoxon's Rank Sum Test — P-value for Percent Change to Week 12. No adjustment for multiplicity was performed
Statistical Analysis 3: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in BAP after 24-week treatment between the two treatment groups; Test type: Superiority or Other; p < 0.001, Wilcoxon's Rank Sum Test — P-value for Percent Change to Week 24. No adjustment for multiplicity was performed
Statistical Analysis 4: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in BAP after 52-week treatment between the two treatment groups; Test type: Superiority or Other; p = 0.060, Wicoxon's Rank Sum Test — P-value for Percent Change to Week 52. No adjustment for multiplicity was performed
Statistical Analysis 5: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in BAP from baseline to the last measurement point between the two treatment groups; Test type: Superiority or Other; p = 0.130, Wilcoxon's Rank Sum Test — P-value for Percent Change to Last Measurement. No adjustment for multiplicity was performed

7. Secondary Outcome: Percent Change in Biochemical Markers of Bone Metabolism - Serum Type I Collagen Crosslinked C-telopeptide (CTX)
Description: Percent change in serum type I collagen crosslinked C-telopeptide (CTX) from baseline to the individual visits and last measurement point.
Time Frame: Baseline to Weeks 4, 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in CTX
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 136 | 67
percent change in CTX
  Percent Change to Week 4 (n=124, n=63) | 2.78 (40.73) | -2.05 (28.17)
  Percent Change to Week 12 (n=121, n=61) | 46.52 (69.52) | -3.56 (27.90)
  Percent Change to Week 24 (n=119, n=59) | 82.27 (110.54) | 4.39 (37.97)
  Percent Change to Week 52 (n=113, n=58) | 84.81 (124.23) | 13.50 (39.47)
  Percent Change to Last Measurement (n=126, n=65) | 79.41 (119.61) | 11.64 (38.61)
Statistical Analysis 1: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in CTX after 4-week treatment between the two treatment groups; Test type: Superiority or Other; p = 0.976, Wilcoxon's Rank Sum Test — P-value for Percent Change to Week 4. No adjustment for multiplicity was performed
Statistical Analysis 2: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in CTX after 12-week treatment between the two treatment groups; Test type: Superiority or Other; p < 0.001, Wilcoxon's Rank Sum Test — P-value for Percent Change to Week 12. No adjustment for multiplicity was performed
Statistical Analysis 3: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in CTX after 24-week treatment between the two treatment groups; Test type: Superiority or Other; p < 0.001, Wilcoxon's Rank Sum Test — P-value for Percent Change to Week 24. No adjustment for multiplicity was performed
Statistical Analysis 4: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in CTX after 52-week treatment between the two treatment groups; Test type: Superiority or Other; p < 0.001, Wilcoxon's Rank Sum Test — P-value for Percent Change to Week 52. No adjustment for multiplicity was performed
Statistical Analysis 5: Comparison: Teriparatide vs Placebo; Null hypothesis: there is no difference in the percent change in CTX from baseline to the last measurement point between the two treatment groups; Test type: Superiority or Other; p < 0.001, Wilcoxon's Rank Sum Test — P-value for Percent Change to Last Measurement. No adjustment for multiplicity was performed

8. Secondary Outcome: Vertebral Fractures by Central X-ray Assessment
Description: Number of vertebral fractures observed from Visit 1 (study entry) through Visit 19 (Week 52). All new or worsened vertebral fractures were defined as a deterioration of at least one grade in a semiquantitative score by X-ray assessment. Number of subjects with fractures and number of fractured vertebra(e) were counted.
Time Frame: Baseline through 52 weeks
Population: Number of randomized participants who received at least one dose of study drug and with at least one post-treatment measurement. The n's are the number of participants with fractures.
Measure: Number; unit: number of fractures
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 136 | 67
number of fractures
  New Fractures (n=5, n=4) | 7 | 5
  Worsening Fractures (n=2, n=0) | 3 | 0

9. Secondary Outcome: Fractures by Investigators Assessment
Description: Vertebral and nonvertebral fractures assessed by the investigator or subinvestigator after starting the study treatment. Traumatic fractures were those caused by falling from above standing height or a high velocity (car) accident. Fractures were assessed to be "fragility" if they occurred without trauma.
Time Frame: Baseline through 52 Weeks
Population: as for outcome 2
Measure: Number; unit: number of fractures
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 136 | 67
number of fractures
  Vertebral Fracture - Fragility | 0 | 1
  Vertebral Fracture - Traumatic | 0 | 0
  Non-Vertebra Fracture - Fragility | 1 | 1
  Non-Vertebra Fracture - Traumatic | 2 | 3

10. Secondary Outcome: Back Pain Severity
Description: Severity of back pain at baseline, individual visits and the last measurement point. Back pain was measured on a scale of 1 (none) to 4 (severe).
Time Frame: Baseline, Weeks 12, 24, 36, 52
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 136 | 67
participants
  Baseline: 1 - None | 77 | 36
  Baseline: 2 - Mild | 47 | 26
  Baseline: 3 - Moderate | 12 | 4
  Baseline: 4 - Severe | 0 | 1
  Week 12: 1 - None | 79 | 41
  Week 12: 2 - Mild | 44 | 18
  Week 12: 3 - Moderate | 8 | 5
  Week 12: 4 - Severe | 0 | 0
  Week 24: 1 - None | 87 | 42
  Week 24: 2 - Mild | 34 | 15
  Week 24: 3 - Moderate | 6 | 4
  Week 24: 4 - Severe | 0 | 0
  Week 36: 1 - None | 82 | 42
  Week 36: 2 - Mild | 36 | 15
  Week 36: 3 - Moderate | 5 | 4
  Week 36: 4 - Severe | 0 | 0
  Week 52: 1 - None | 84 | 42
  Week 52: 2 - Mild | 32 | 12
  Week 52: 3 - Moderate | 5 | 5
  Week 52: 4 - Severe | 0 | 1
  Last Measurement: 1 - None | 90 | 44
  Last Measurement: 2 - Mild | 36 | 14
  Last Measurement: 3 - Moderate | 5 | 5
  Last Measurement: 4 - Severe | 0 | 1

11. Secondary Outcome: Percent Change in Bone Mineral Density at Lumbar Spine (L2-L4) During Open Label Phases at 76 Weeks and 104 Weeks
Description: Percent change in bone mineral density (BMD) at lumbar spine (L2-L4) from baseline to the last measurement point.
Time Frame: Baseline, 76 Weeks, 104 Weeks
Population: Number of randomized participants with at least one dose of study drug and at least one post-treatment measurement.
Measure: Mean (Standard Deviation); unit: percent change in BMD
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 131 | 63
percent change in BMD
  Percent Change to Week 76; n=113, n=55 | 11.93 (5.79) | 6.39 (4.74)
  Percent Change to Week 104; n=92, n=47 | 13.42 (6.12) | 9.11 (5.14)

12. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) at Lumbar Spine (L1-L4) During Open Label Phases at 76 Weeks and 104 Weeks
Description: Percent change in bone mineral density at lumbar spine (L1-L4) from baseline to the last measurement point.
Time Frame: Baseline, 76 Weeks, 104 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in BMD
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 131 | 63
percent change in BMD
  Percent Change to Week 76; n=113, n=55 | 12.24 (5.86) | 6.63 (4.69)
  Percent Change to Week 104; n=92, n=47 | 14.01 (6.41) | 9.46 (5.35)

13. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) at Total Hip During Open Label Phases at 76 Weeks and 104 Weeks
Description: Percent change in bone mineral density (BMD) at total hip from baseline to the last measurement point.
Time Frame: Baseline, 76 Weeks, 104 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in BMD
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 130 | 62
percent change in BMD
  Percent Change to Week 76; n=112, n=54 | 3.02 (3.79) | 1.64 (4.63)
  Percent Change to Week 104; n=91, n=46 | 3.67 (3.98) | 2.46 (3.54)

14. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) at Femoral Neck During Open Label Phases at 76 Weeks and 104 Weeks
Description: Percent change in bone mineral density at femoral neck from baseline to the last measurement point.
Time Frame: Baseline, 76 Weeks, 104 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in BMD
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 130 | 62
percent change in BMD
  Percent Change to Week 76; n=112, n=54 | 2.68 (4.45) | 1.17 (4.81)
  Percent Change to Week 104; n=91, n=46 | 3.26 (4.25) | 2.19 (4.81)

15. Secondary Outcome: Percent Change in Biochemical Markers of Bone Metabolism - Serum Procollagen I N-terminal Propeptide (PINP) During Open Label Phases at 76 Weeks and 104 Weeks
Description: as for outcome 5
Time Frame: Baseline, 76 Weeks, 104 Weeks
Population: Number of randomized participants with at least one dose of study drug and with at least one post-treatment measurement.
Measure: Mean (Standard Deviation); unit: percent change in PINP
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 136 | 67
percent change in PINP
  Percent change to Week 76; n=113, n=55 | 115.45 (174.07) | 97.28 (131.64)
  Percent change to Week 104; n=92, n=47 | 74.71 (112.48) | 134.89 (180.76)

16. Secondary Outcome: Percent Change in Biochemical Markers of Bone Metabolism - Serum Bone-specific Alkaline Phosphatase (BAP) During Open Label Phases at 76 Weeks and 104 Weeks
Description: as for outcome 6
Time Frame: Baseline, 76 Weeks, 104 Weeks
Population: Number of randomized participants with at least one dose of study drug and with at least one post-treatment measurement.
Measure: Mean (Standard Deviation); unit: percent change in BAP
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 136 | 67
percent change in BAP
  Percent Change to Week 76; n=113, n=55 | 17.49 (66.40) | 15.71 (64.96)
  Percent Change to Week 104; n=92, n=47 | -1.52 (54.38) | 16.45 (71.72)

17. Secondary Outcome: Percent Change in Biochemical Markers of Bone Metabolism - Serum Type I Collagen Crosslinked C-telopeptide (CTX) During Open Label Phases at 76 Weeks and 104 Weeks
Description: Percent change in serum type I collagen crosslinked C-telepeptide (CTX) from baseline to the individual visits and last measurement point.
Time Frame: Baseline, 76 Weeks, 104 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in CTX
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 136 | 67
percent change in CTX
  Percent Change to Week 76; n=104, n=53 | 85.85 (137.13) | 86.98 (132.81)
  Percent Change to Week 104; n=85, n=45 | 54.39 (111.97) | 72.84 (100.91)

18. Secondary Outcome: Vertebral Fractures by Central X-ray Assessment During Entire Study Period of 104 Weeks
Description: Number of vertebral fractures observed from Visit 1 (study entry) through 104 weeks. All new or worsened vertebral fractures were defined as a deterioration of at least one grade in a semiquantitative score by X-ray assessment. Number of subjects with fractures and number of fractured vertebra(e) were counted.
Time Frame: Baseline through 104 Weeks
Population: Number of randomized participants who received at least one dose of study drug and with at least on post-treatment measurement. The n's are the number of participants with fractures.
Measure: Number; unit: number of fractures
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 136 | 67
number of fractures
  New Fractures at 104 Weeks (n=5, n=6) | 7 | 7
  Worsening Fractures at 104 Weeks (n=2, n=2) | 3 | 3

19. Secondary Outcome: Fractures by Investigators Assessment During Entire Study Period of 104 Weeks
Description: as for outcome 9
Time Frame: Baseline Through 104 Weeks
Population: as for outcome 2
Measure: Number; unit: number of fractures
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 136 | 67
number of fractures
  Vertebral Fracture - Fragility - 104 Weeks | 0 | 1
  Vertebral Fracture - Traumatic - 104 Weeks | 0 | 0
  Non-Vertebra Fracture - Fragility - 104 Weeks | 1 | 1
  Non-Vertebra Fracture - Traumatic - 104 Weeks | 3 | 4

20. Secondary Outcome: Back Pain Severity During Open Label Phases at 76 Weeks and 104 Weeks
Description: Severity of back pain at 76 weeks and 104 weeks. Back pain was measured on a scale of 1 (none) to 4 (severe).
Time Frame: Baseline, 76 Weeks, 104 Weeks
Population: Number of randomized participants who received at least one dose of study drug and with at least on post-treatment measurement.
Measure: Number; unit: participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 136 | 67
participants
  Week 76: 1- None | 78 | 38
  Week 76: 2- Mild | 31 | 13
  Week 76: 3- Moderate | 4 | 4
  Week 76: 4- Severe | 0 | 0
  Week 104: 1- None | 66 | 32
  Week 104: 2- Mild | 23 | 13
  Week 104: 3- Moderate | 3 | 2
  Week 104: 4- Severe | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and Other Adverse Events are reported for both treatment arms for the following time frames: double-blind treatment (During 52 weeks); open-label treatment (During 76 weeks); open-label treatment (During 104 weeks).
Groups:
- Teriparatide (During 52 Weeks); Teriparatide (During 76 Weeks); Teriparatide (During 104 Weeks): 20 micrograms for 104 weeks
- Placebo (During 52 Weeks); Placebo (During 76 Weeks); Placebo (During 104 Weeks): Placebo for 52 weeks. After 52 weeks, all patients on placebo can receive 20 micrograms teriparatide for 52 weeks
Arm/Group | Teriparatide (During 52 Weeks) | Placebo (During 52 Weeks) | Teriparatide (During 76 Weeks) | Placebo (During 76 Weeks) | Teriparatide (During 104 Weeks) | Placebo (During 104 Weeks)
Serious Adverse Events (participants affected / at risk) | 7/136 | 7/67 | 10/136 | 9/67 | 12/136 | 13/67
Other Adverse Events (participants affected / at risk) | 115/136 | 59/67 | 123/136 | 60/67 | 125/136 | 64/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (During 52 Weeks) (N=136) | Placebo (During 52 Weeks) (N=67) | Teriparatide (During 76 Weeks) (N=136) | Placebo (During 76 Weeks) (N=67) | Teriparatide (During 104 Weeks) (N=136) | Placebo (During 104 Weeks) (N=67)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Artery dissection (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (During 52 Weeks) (N=136) | Placebo (During 52 Weeks) (N=67) | Teriparatide (During 76 Weeks) (N=136) | Placebo (During 76 Weeks) (N=67) | Teriparatide (During 104 Weeks) (N=136) | Placebo (During 104 Weeks) (N=67)
Constipation (Gastrointestinal disorders) | 10 (11) | 2 (3) | 11 (13) | 4 (5) | 12 (14) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 0 (0) | 7 (11) | 4 (4) | 8 (15) | 6 (7)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 6 (7) | 2 (2) | 7 (8) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 6 (6) | 4 (6) | 7 (7) | 5 (7)
Injection site reaction (General disorders) | 5 (7) | 8 (14) | 5 (7) | 8 (14) | 5 (7) | 8 (14)
Seasonal allergy (Immune system disorders) | 8 (8) | 4 (4) | 8 (8) | 5 (5) | 12 (15) | 6 (8)
Cystitis (Infections and infestations) | 7 (8) | 2 (2) | 7 (10) | 4 (4) | 8 (11) | 4 (4)
Nasopharyngitis (Infections and infestations) | 38 (66) | 27 (37) | 45 (89) | 29 (51) | 55 (113) | 32 (68)
Contusion (Injury, poisoning and procedural complications) | 8 (10) | 4 (4) | 11 (13) | 5 (5) | 14 (16) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 9 (9) | 6 (7) | 11 (12) | 7 (8) | 14 (15) | 11 (12)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 2 (2) | 4 (4) | 2 (2) | 5 (5) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 4 (5) | 8 (9) | 7 (9) | 10 (11) | 9 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (18) | 9 (11) | 22 (24) | 15 (20) | 25 (33) | 16 (23)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2) | 5 (6) | 1 (2) | 8 (9) | 2 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (10) | 4 (4) | 10 (11) | 5 (5) | 14 (16) | 6 (6)
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 5 (6) | 4 (4) | 7 (8) | 5 (5)
Dizziness (Nervous system disorders) | 8 (10) | 3 (3) | 11 (14) | 3 (4) | 12 (18) | 5 (7)
Headache (Nervous system disorders) | 9 (11) | 3 (3) | 10 (14) | 4 (5) | 10 (15) | 4 (5)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 7 (7) | 2 (2) | 8 (9) | 3 (3)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 3 (3) | 9 (16) | 3 (4) | 10 (22) | 3 (6)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (5) | 7 (7) | 4 (5) | 7 (7) | 4 (5)
Eczema (Skin and subcutaneous tissue disorders) | 5 (6) | 5 (5) | 6 (7) | 5 (6) | 6 (7) | 5 (6)
Dental care (Surgical and medical procedures) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 7 (10) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 4 (5) | 0 (0) | 5 (7) | 1 (1) | 7 (11) | 4 (4)

LIMITATIONS AND CAVEATS:
Original data presented were for the 52-week double-blinded treatment phase; results of the open label phases at 76 weeks and 104 weeks have now been added

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days